CLINICAL TRIAL: NCT00254358
Title: A Brain Imaging Study of Nicotine Release in Cigarette Smokers
Status: Terminated | Type: Observational
Why Stopped: It was decided to use a different protocol with a different radioligand
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Herzog Hospital (Other)
Responsible Party: Dr. Aviv Weinstein, Hadassah Medical Organization
Other Study IDs: 842902-HMO-CTIL
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Nicotine Dependence
Keywords: Nicotine; Dopamine; IBZM
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Tobacco Smoking is the most prevalent addiction in society today causing directly major health hazards and sharing morbidity with other psychiatric disorders. Nicotine binds to acetylcholine receptors and thus elevates DA release and inhibits DA transport. There are few studies using advanced brain imaging techniques to investigate how nicotine releases dopamine in humans. These studies utilized dopamine displacement paradigms with [11C] Raclopride binding to D2 receptor in Positron Emission Tomography (PET). There is evidence that smokers (particularly those who enjoyed smoking) showed decreased [11C] Raclopride binding in the caudate/nucleus accumbens and putamen after smoking cigarettes. These results also indicated that the effects of nicotine on dopaminergic neurotransmission are mediated by pleasure and craving. We propose to investigate the effects of smoking a cigarette ad lib on dopamine release by using dopamine competition paradigm with [I123] IBZM in SPECT. Secondly, we will test the hypothesis that dopamine deficiency is a major vulnerability factor for smoking. This may provide further evidence that dopamine deficiency in some smokers pre-disposes them to enjoy and desire smoking cigarettes more than others.

ELIGIBILITY:
Inclusion Criteria:

* Chronic smokers and healthy non-smokers.

Exclusion Criteria:

* Pregnant and breast feeding women.
* Age below 20.
* Neurological disorders.
* Others drugs.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: smokers in treatment with bupropion
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-04; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yodphat Krausz, MD, Principal Investigator — Hadassah Medical Organization